CLINICAL TRIAL: NCT06445439
Title: Optimal Pacing Rate for Cardiac Resynchronization Therapy After Atrioventricular Node Ablation in Persistent Atrial Fibrillation and Heart Failure
Brief Title: Optimal Pacing Rate for Cardiac Resynchronization Therapy
Acronym: OPT-RATE AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00006952
Record Dates: First submitted 2024-03-25; First posted 2024-06-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign half of the participants to a starting rate of 60 bpm and then switch them to a rate of 80 bpm for 3 months, and vice versa.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 60 bpm, then 80 bpm (Experimental): Pacing rate of 60 bpm for the first 3 months, then switch to 80 bpm for the next 3 months.
  Interventions: Device: Pacing rate of 80 bpm; Device: Pacing rate of 60 bpm
- 80 bpm, then 60 bpm (Experimental): Pacing rate of 80 bpm for the first 3 months, then switch to 60 bpm for the next 3 months.
  Interventions: Device: Pacing rate of 80 bpm; Device: Pacing rate of 60 bpm

INTERVENTIONS:
Device: Pacing rate of 80 bpm — Pacing rate of 80 bpm
Device: Pacing rate of 60 bpm — Pacing rate of 60 bpm

SUMMARY:
This is a prospective, randomized crossover study. The objective of the study is to determine if a pacing rate of 80 beats per minute (bpm) improves exercise tolerance during the 6-minute walk test. The investigators will randomly assign half of the participants to a starting rate of 60 bpm and then switch them to a rate of 80 bpm for 3 months, and vice versa.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) after atrioventricular node (AVN) ablation for permanent atrial fibrillation (AF) has led to better outcomes in heart failure (HF) patients with reduced ejection fraction (HFrEF) and with preserved ejection fraction (HFpEF) compared to pharmacotherapy. Emerging evidence has demonstrated patients with HFpEF may benefit from a higher heart rate compared to standard heart-lowering therapies. The optimal pacing rate for CRT after AVN ablation in persistent AF and HFpEF remains unknown.

This is a prospective, randomized crossover study. The objective of the study is to determine if a pacing rate of 80 beats per minute (bpm) improves exercise tolerance during the 6-minute walk test.

The investigators will randomly assign half of the participants to a starting rate of 60 bpm and then switch them to a rate of 80 bpm for 3 months, and vice versa. Patient mortality and HF hospitalizations will be recorded at each phase. An electrocardiogram, echocardiogram, pacemaker interrogation, BNP and creatinine levels, KCCQ-12, six-minute walk test, and physical activity measure will be obtained at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. History of persistent or permanent atrial fibrillation
3. Implantation of CRT or conduction system pacing in prior 3 months to 5 years of study start
4. History of intrinsic AVN block or have undergone AVN ablation in prior 3 months to 5 years of study start
5. LVEF ≥ 50%
6. N-terminal pro-B-type natriuretic peptide (NT-proBNP) >400 pg/mL in the last 24 months
7. Clinical HF diagnosis or NYHA class II or higher
8. Able to provide informed consent

Exclusion Criteria:

1. LVEF <50%
2. Wide QRS (greater than 150ms)
3. Isolated RV pacing
4. Severe valvular disease
5. Severe coronary artery disease as defined by one of the following:

   1. ACS or PCI within 1 year
   2. Any angina (CCS class 1+)
   3. Unrevascularizable severe CAD (>70% stenosis in 1+ major vessels and/or based on functional assessment)
6. ESRD
7. Significant primary pulmonary disease on home oxygen
8. Major orthopedic issues, such as being wheelchair bound and/or unable to perform a six-minute walk test
9. Ventricular ectopy >15% premature ventricular contractions (PVC)
10. End stage cancer diagnosis
11. Life expectancy less than one year
12. Palliative or hospice care
13. Hypertrophic cardiomyopathy (HCM)
14. Uncorrected ventricular septal defect
15. Infiltrative cardiomyopathy (CM)
16. Uncontrolled hypertension as defined by blood pressure >160/100 mm Hg on two measurements ≥15 minutes apart
17. Hemoglobin <7 g/dL
18. Age >90 years old
19. Pregnant or intends to become pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance as measured by the Six-Minute Walk Test | 3 months
  Exercise tolerance as measured by the Six-Minute Walk Test

SECONDARY OUTCOMES:
Quality of life as measured by the Kansas City Cardiomyopathy Questionnaire | 3 months
  Quality of life as measured by the Kansas City Cardiomyopathy Questionnaire
Function as measured by the International Physical Activity Questionnaire | 3 months
  Function as measured by the International Physical Activity Questionnaire
Change in B-type natriuretic peptide (BNP) | 3 months
  Change in B-type natriuretic peptide (BNP)
Change in creatinine | 3 months
  Change in creatinine
Change in New York Heart Association Class | 3 months
  Change in New York Heart Association Class
Atrial fibrillation burden | 3 months
  Atrial fibrillation burden as measured by pacemaker
Hospitalization for heart failure | 3 months
  Hospitalization for heart failure
Death due to heart failure | 3 months
  Death due to heart failure
Death due to myocardial infarction | 3 months
  Death due to myocardial infarction
Death due to stroke | 3 months
  Death due to stroke
Hospitalization for atrial fibrillation | 3 months
  Hospitalization for atrial fibrillation
Administration of loop diuretic/anti-arrhythmic drug | 3 months
  Administration of loop diuretic/anti-arrhythmic drug

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Thomaides, MD, Principal Investigator — MedStar Health
Locations (5):
- United States (5):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Southern Maryland Hospital, Clinton, Maryland
  - MedStar Heart and Vascular Office at Fairfax, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Study data available from PI upon request.